CLINICAL TRIAL: NCT02354651
Title: Response to Diaphragmatic Pacing in Subjects With Pompe Disease
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201600161-N; 003-2013 (Other: University of Florida pre-conversion); 1R21HD090752-01 (NIH)
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pompe Disease
Keywords: Pompe disease; mechanical ventilation; diaphragm pacing
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients With Pompe Disease Eligible for Diaphragm Pacing: Patients will receive tests of breathing pattern, phrenic nerve stimulation, maximal inspiratory pressure (MIP), forced expiration, and EMG.
  Interventions: Other: Diaphragm conditioning via phrenic nerve stimulation

INTERVENTIONS:
Other: Diaphragm conditioning via phrenic nerve stimulation — Diaphragm pacing will be prescribed by the patient's clinical team.

SUMMARY:
The purpose of this study is to determine the effect of diaphragm pacing on respiratory function in subjects with Pompe disease by evaluating the duration and pattern of spontaneous respiratory function versus paced ventilation respiratory function in patients with Pompe disease who have received the NeuDx Diaphragm pacer (DPS).

DETAILED DESCRIPTION:
Subjects with Pompe disease who are scheduled to receive a NeuRx Diaphragm pacer (DPS) will be invited to participate in this study. The following tests will be performed during participation in the study:

1. Forced expiratory tests
2. Maximal Inspiratory Pressure (MIP)
3. Resting Breathing Pattern
4. Phrenic Nerve Function Evaluation with EMG
5. Severe Respiratory Insufficiency Questionnaire
6. Magnetic stimulation
7. Diaphragm conditioning consisting of:

   1. The external stimulator settings
   2. The duration of diaphragm stimulation
   3. Off-ventilator spontaneous breathing (SB)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pompe disease as defined by mutational analysis, GAA enzyme activity assay in blood spot, and/or fibroblast culture less than 40% of control value
* Medically and functionally eligible for NeuRx DPS implantation, as determined by a clinical surgical evaluation. The surgeon will determine eligibility through pulmonary function tests, ability to stimulate your diaphragm, and arterial blood gas levels. Eligibility may also be determined by your response to traditional respiratory strengthening exercises without a pacemaker.
* History of mechanical ventilation dependence (six or more hours of invasive or non-invasive mechanical ventilation support daily for at least 21 days in duration

Exclusion Criteria:

* Current participation in another treatment study (other than enzyme replacement therapy) directed at improving diaphragm function
* Unable to complete pulmonary function testing

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Pompe disease who are eligible for NeuRx DPS implantation
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2022-06 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Smith, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were eligible to receive a diaphragmatic pacemaker as part of their clinical care. Some subjects who enrolled decided not to include pacing as part of their clinical care (n=2), or were found to have medical conditions that made them ineligible (n=1).
Groups:
- Patients With Pompe Disease Eligible for Diaphragm Pacing: Patients will receive tests of breathing pattern, phrenic nerve stimulation, maximal inspiratory pressure (MIP), forced expiration, and EMG.
  Diaphragm conditioning via phrenic nerve stimulation: Diaphragm conditioning will be prescribed by the patient's clinical team.
Period: Overall Study
Arm/Group | Patients With Pompe Disease Eligible for Diaphragm Pacing
Started | 9
Completed | 6
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants who underwent implantation of a diaphragm pacing system.
Groups:
- Pompe Subjects Receiving NeuDx DPS: Patients will receive resting breathing pattern evaluation, phrenic nerve stimulation, maximal inspiratory pressure (MIP) testing, forced expiratory testing, and EMG.
  Diaphragm conditioning via phrenic nerve stimulation: Diaphragm pacing will be prescribed by the patient's clinical team.
Arm/Group | Pompe Subjects Receiving NeuDx DPS
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.5 [3 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Ventilator-Free Breathing [Mean (Full Range); unit: hours of unassisted ventilation per day] — Hours of daily ventilation unassisted by positive pressure ventilation.
  hours of unassisted ventilation per day | 0.52 [0 to 1.5]

OUTCOME MEASURES:

1. Primary Outcome: Off-ventilator Spontaneous Breathing (SB) at Baseline and Day 180
Description: The patient will undergo an initial trial of unassisted breathing with the diaphragm pacer turned on. The duration of SB with pacing will be increased to tolerance, using a protocol. If the patient cannot initially complete at least 30-minute bouts of paced SB, then the focus of breathing trials will be to breathe with reduced support from the mechanical ventilator. These measures were generated utilizing ventilator chip data for SB that has been averaged.
Time Frame: Baseline, Day 180
Population: Full sample
Measure: Mean (Full Range); unit: hours per day
Groups:
- Pompe Subjects Receiving NeuRx DPS: Patients will receive resting breathing pattern evaluation, phrenic nerve stimulation, maximal inspiratory pressure (MIP) testing, forced expiratory testing, and EMG.
  Diaphragm conditioning via phrenic nerve stimulation: Diaphragm pacing will be prescribed by the patient's clinical team.
Arm/Group | Pompe Subjects Receiving NeuRx DPS
Number analyzed (Participants) | 6
hours per day
  Baseline | 0.52 [0 to 1.5]
  Day 180 | 4.72 [.04 to 12]

2. Secondary Outcome: Maximal Inspiratory Pressure (MIP) at Baseline and Day 180
Description: MIP will be measured with a manometer connected to the airway opening of the subject, which occludes the airway and prevents airflow. A nose clip will be used to prevent leakage and the subject is instructed to suck air from the tube with as much force as possible. Measurements will be obtained with the subject sitting upright. Transdiaphragmatic pressure (Pdi) may be calculated with esophageal and gastric manometry during MIP. The measurement will be taken three times and the best value will be reported.
Time Frame: Baseline, Day 180
Population: Subjects 4 and 6 were unavailable for MIP testing at baseline; Subjects 1 and 3 were unavailable for MIP testing at 6 months.
Measure: Mean (Full Range); unit: cm H2O
Arm/Group | Pompe Subjects Receiving NeuRx DPS
Number analyzed (Participants) | 4
cm H2O
  Baseline | 35.6 [12.8 to 65]
  180 Days | 32.7 [8.3 to 61]

3. Secondary Outcome: Change in Resting Breathing Pattern
Description: Resting ventilatory flow and timing will be recorded with a pneumotachograph and pressure transducer connected to the airway opening, to calculate minute ventilation. If a patient routinely uses MV throughout the day, the sensing equipment can be placed in series to the breathing tubes. Breathing pattern will be measured for a minimum of ten minutes.
Time Frame: Day 180
Population: Minute ventilation during off-ventilator breathing was assessed with and without diaphragm pacing at approximately 6 months post-implant.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Pompe Subjects Receiving NeuRx DPS
Number analyzed (Participants) | 4
L/min
  Without diaphragm pacer | 5.05 (1.73)
  With diaphragm pacer | 5.41 (3.54)

4. Secondary Outcome: Diaphragm Electromyogram (EMG) at Day 180
Description: This activity reflects the activity of the diaphragm and phrenic nerve. The wires that are implanted for diaphragm pacemaker will be connected to a computer and recording equipment to monitor the activity of the diaphragm muscle during breathing at the lowest level of ventilator assistance. This EMG data is measured in units of microvolts per second and expressed as a percentage of the level of diaphragm EMG activity recorded during MIP maneuvers.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: RMS diaphragm (% of MIP)
Arm/Group | Pompe Subjects Receiving NeuRx DPS
Number analyzed (Participants) | 4
RMS diaphragm (% of MIP) | 57.3 (38.9)

5. Other Pre Specified Outcome: Hours Per Day of Diaphragm Pacing
Description: Number of hours used per day diaphragm pacing occurred by subjects
Time Frame: 180 days
Population: Patients with Pompe disease who received diaphragm pacing
Measure: Mean (Full Range); unit: hours per day of diaphragm pacing
Arm/Group | Patients With Pompe Disease Eligible for Diaphragm Pacing
Number analyzed (Participants) | 6
hours per day of diaphragm pacing | 20.3 [2 to 24]

6. Other Pre Specified Outcome: Magnetic Stimulation
Description: EMG response to supramaximal bilateral stimulation of the phrenic nerves.
Time Frame: 180 Days
Population: Magnetic stimulation was used as assessment for determining clinical eligibility for diaphragm pacing. It was not available at follow-up observational visits.
Arm/Group | Patients With Pompe Disease Eligible for Diaphragm Pacing
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Severe Respiratory Insufficiency Questionnaire
Description: Patient reported measure of impact of respiratory insufficiency on functional mobility
Time Frame: 180 days
Population: The Severe Respiratory Insufficiency Questionnaire was validated only in adults. Adults who participated did not complete the questionnaire at Day 180.
Arm/Group | Patients With Pompe Disease Eligible for Diaphragm Pacing
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Forced Expiratory Flow
Description: Peak expiratory flow obtained during voluntary cough
Time Frame: 180 days
Population: Only 2 patients were able to complete voluntary cough during a 180-day visit
Measure: Mean (Full Range); unit: L/min
Arm/Group | Pompe Subjects Receiving NeuDx DPS
Number analyzed (Participants) | 2
L/min | 42.65 [36.4 to 48.9]

ADVERSE EVENTS:
Time Frame: Longitudinal observational data through January 2019. Post-operative observation time frame ranged from 89 months in subject 1, to 45 months in subject 6..
Arm/Group | Pompe Subjects Receiving NeuRx DPS
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pompe Subjects Receiving NeuRx DPS (N=6)
Scoliosis requiring spinal fusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizures (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pompe Subjects Receiving NeuRx DPS (N=6)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Occipital pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Damaged infusion port (Product Issues) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Breakage of pacemaker external wires (Product Issues) | 5 (9)

LIMITATIONS AND CAVEATS:
This was a pilot observational study that tracked an unusual clinical intervention in a rare disease; thus, generalizability is difficult to ascertain. Consistent measurement times were difficult to access some patients who resided great distances from the study center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT02354651/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02354651/SAP_001.pdf